CLINICAL TRIAL: NCT01721187
Title: Functional Magnetic Resonance Imaging Study of the Valuation of Food as a Function of Satiety
Brief Title: Satiety Effects on the Neural Valuation of Food
Status: Completed | Type: Observational
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: Institute for Human Development and Potential (IHDP), Singapore (Other)
Responsible Party: Principal Investigator, MChee, Professor, Duke-NUS Graduate Medical School
Other Study IDs: VOFIO3G
Record Dates: First submitted 2012-10-23; First posted 2012-11-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Fasting; Fed
Keywords: fMRI; Satiety; Willingness to Pay; Incentive Delay; Dietary Disinhibition
MeSH Terms: conditions — Fasting; Lecithin Cholesterol Acyltransferase Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — (NA)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low disinhibition: fMRI during fed and fasted states
- High disinhibition: fMRI during fed and fasted states

SUMMARY:
Using fMRI, this study will explore the neural correlates of satiety when individuals make decisions about food. The investigators will also examine individual differences in satiety effects.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity
* 21 to 45 years old
* English as first language
* Right-handed
* Have normal eyesight, or have long-sightedness or myopia within +8.0 to -8.0 diopters (unless corrected by contact lenses)
* Weigh less than 100kg with an abdominal circumference of less than 120cm
* Non-smoker, or only smoke occasionally (less than 5 sticks a week)
* Consume less than 2 units (200 mg) of caffeine a day
* Consume less than 21 units of alcohol per week (e.g. 500ml 5% beer = 2.5 units, 250ml 14% wine = 3.5 unit)
* Habitually sleep before 1am and wake before 9am

Exclusion Criteria:

* On a restrictive diet (e.g., vegetarian/vegan diet)
* History of food allergies
* History of psychiatric or neurological disorders
* History of chronic medical illness
* Metal implants in or on the body (e.g. braces, dental retainers, pacemakers)
* Shift worker
* Claustrophobic
* High astigmatism (high = >2.00 diopters)
* Colour-blind

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
fMRI - Willingness to Pay task (BDM auction) | Fed and fasted visits (Wks 1 & 2)
  A measurement of how much participants are willing to pay for foods and non-foods, as an assay for subjective value of goods.
fMRI - Monetary and Food Incentive Delay task | Fed and fasted visits (Wks 1 & 2)
  A measurement of neural response to anticipating and receiving money and food rewards.

CONTACTS AND LOCATIONS:
Overall Officials: Michael WL Chee, MBBS, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Centre for Cognitive Neuroscience scanner suite, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Plassmann H, O'Doherty J, Rangel A. Orbitofrontal cortex encodes willingness to pay in everyday economic transactions. J Neurosci. 2007 Sep 12;27(37):9984-8. doi: 10.1523/JNEUROSCI.2131-07.2007. PMID 17855612
- [Background] Knutson B, Westdorp A, Kaiser E, Hommer D. FMRI visualization of brain activity during a monetary incentive delay task. Neuroimage. 2000 Jul;12(1):20-7. doi: 10.1006/nimg.2000.0593. PMID 10875899